CLINICAL TRIAL: NCT05241275
Title: XENON ILD: 129Xe MRI to Evaluate aNtifibrotic respOnse and progressioN in ILD
Brief Title: Xenon MRI and Progressive ILD
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Principal Investigator, Bastiaan Driehuys, Professor of Radiology, Duke University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00109322
Record Dates: First submitted 2022-02-03; First posted 2022-02-15 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Idiopathic Pulmonary Fibrosis; Progressive Pulmonary Fibrosis
Keywords: Magnetic Resonance Imaging
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Progressive Pulmonary Fibrosis (Experimental): Whether magnetic resonance imaging (MRI) using inhaled hyper-polarized 129 Xenon gas can help visualize impaired lung function to detect changes over time in Progressive Pulmonary Fibrosis patients receiving approved treatments.
  Interventions: Drug: Hyperpolarized 129 Xenon Gas Comparing Progressive Pulmonary Fibrosis Treatment

INTERVENTIONS:
Drug: Hyperpolarized 129 Xenon Gas Comparing Progressive Pulmonary Fibrosis Treatment — Whether magnetic resonance imaging (MRI) using inhaled hyper-polarized 129 Xenon gas can help visualize impaired lung function to detect changes over time in Progressive Pulmonary Fibrosis

SUMMARY:
The XENON ILD study is a single arm, un-blinded study at Duke University enrolling patients with non-idiopathic pulmonary fibrosis (IPF) progressive fibrosis (PF) interstitial lung disease (ILD). Patients who meet criteria for ILD-progression (defined below in inclusion/exclusion criteria) will be consented prior to the initiation of anti-fibrotic therapy. Subjects will undergo an approximately hour long comprehensive MRI protocol, including administration of multiple doses of hyperpolarized 129Xe. The subjects will have this initial study prior to initiation of anti-fibrotic therapies and repeat MRI studies at 3, 6 and 12 months following the initiation of therapy. If subjects do not decide to initiate anti-fibrotic therapy per discussion with their physician, then the 3, 6 and 12 months repeat studies will initiate based on time after enrollment.

DETAILED DESCRIPTION:
The XENON ILD study is a single arm, un-blinded study at Duke University enrolling patients with non-IPF PF-ILD. Patients who meet criteria for ILD-progression (defined below in inclusion/exclusion criteria) will be consented prior to the initiation of anti-fibrotic therapy. Subjects will undergo an approximately hour long comprehensive MRI protocol, including administration of multiple doses of hyperpolarized 129Xe. The subjects will have this initial study prior to initiation of anti-fibrotic therapies and repeat MRI studies at 3, 6 and 12 months following the initiation of therapy. If subjects do not decide to initiate anti-fibrotic therapy per discussion with their physician, then the 3, 6 and 12 months repeat studies will initiate based on time after enrollment. We plan to consent 75 subjects with PF-ILD who are candidates for anti-fibrotic therapy to slow ILD progression. We will ensure that the study will include at least 38 subjects who start anti-fibrotic therapy after baseline first MRI scan and continue the therapy until his/her 3 month repeat MRI scan. This will be obtained by a pre-specified increase in the number of subjects until the 38 subject criteria is completed. Subject will not be excluded from the study due to stopping anti-fibrotic therapy for any reason during the study.

Additional studies including pulmonary function studies, plasma and serum for biomarkers, whole blood for DNA (baseline visit only), whole blood for RNA, exhaled breath for biomarkers, 6 minute walk distance and a HRCT (only at the screening visit, 6 month visit, and 12 month visit) will be performed to determine how 129Xe MRI performs relative to standard of care evaluations for PF-ILD patients. Finally, following the study visits the research team will prospectively follow the patients' clinical course through periodic reviews of the medical record.

ELIGIBILITY:
Inclusion Criteria:

* We will include all patients who are over 18 years of age with a physician-diagnosed ILD of one of the below subtypes based on multidisciplinary consensus

  1. Chronic hypersensitivity pneumonitis
  2. Autoimmune interstitial lung disease (including rheumatoid arthritis-ILD, mixed connective tissue disorder related ILD, myositis related ILD, scleroderma related ILD, and idiopathic pneumonia with autoimmune features)
  3. Idiopathic NSIP
  4. Unclassifiable idiopathic interstitial pneumonia
* Fibrotic lung disease affecting more than 10% of lung volume on high-resolution CT, per Duke radiology review
* Evidence of any of the following criteria for progression of ILD within the 24 months before screening:

  1. Relative decline in FVC % predicted of at least 10%
  2. Relative decline in FVC % predicted ≥ 5% - < 10 combined with either increasing extent of fibrotic changes on HRCT or worsening of respiratory symptoms
  3. Worsening respiratory symptoms and increased extent of fibrosis on HRCT
* Willing and able to give informed consent and adhere to visit/protocol schedules
* Immunosuppressive medication, including azathioprine, cyclosporine, mycophenolate mofetil, rituximab, cyclophosphamide, or oral glucocorticoids are permitted at the discretion of the treating physician

Exclusion Criteria:

* Subject is less than 18 years of age
* Prior treatment with nintedanib or pirfenidone
* Subject is pregnant or lactating
* Prior investigational drug use within 28 days
* MRI is contraindicated based on responses to MRI screening questionnaire
* Respiratory illness of a bacterial or viral etiology within 30 days of MRI
* Acute exacerbation within 30 days of MRI, defined by acute increases in oxygen requirement, bilateral alveolar filling opacities on imaging, and the need for antibiotics and/or systemic steroids
* Subject does not fit into 129Xe vest coil used for MRI
* Subject with ventricular cardiac arrhythmia in the past 30 days.
* Subject has history of cardiac arrest within the last year
* Subject deemed unlikely to be able to comply with instructions during imaging
* Medical or psychological conditions which, in the opinion of the investigator, might create undue risk to the subject or interfere with the subject's ability to comply with the protocol requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-07-19 (Actual); Primary Completion 2025-11-03 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in 129Xe MRI barrier uptake 3 months after anti-fibrotic initiation | Baseline, 3 months
  The outcome will assess changes in 129Xe MRI barrier uptake 3 months after nintedanib initiation.

SECONDARY OUTCOMES:
Change in 129Xe MRI barrier uptake 6 months after anti-fibrotic initiation | Baseline and 6 months
  The outcome will assess changes in 129Xe MRI barrier uptake 6 months after nintedanib initiation.
Change in 129Xe MRI RBC to barrier ratio 3 months after anti-fibrotic initiation | Baseline and 3 months
  RBC to barrier ratio is a ratio of the RBC transfer and barrier values and is reported as a single value
Change in 129Xe MRI RBC to barrier ratio 6 months after anti-fibrotic initiation | Baseline and 6 months
  RBC to barrier ratio is a ratio of the RBC transfer and barrier values and is reported as a single value
Time to disease progression (occurrence of a ≥ 10% drop in percent predicted FVC, all cause death, or lung transplant) in individuals with elevated barrier uptake at baseline greater than 2 standard deviations of a healthy reference cohort | Up to 12 months
  Time to disease progression will be recorded in months
Time to disease progression (occurrence of a ≥ 10% drop in percent predicted FVC, all cause death, or lung transplant) in individuals with decreased RBC transfer at baseline, lower than 2 standard deviations of a healthy reference cohort | Up to 12 months
  Time to disease progression will be recorded in months
Time to disease progression (occurrence of a ≥ 10% drop in percent predicted FVC, all cause death, or lung transplant) in individuals with a reduced RBC to barrier ratio, greater than 2 standard deviations of a healthy reference cohort | Up to 12 months
  RBC to barrier ratio is a ratio of the RBC transfer and barrier values and is reported as a single value. Time to disease progression will be recorded in months
Time to acute exacerbation or respiratory hospitalization in individuals with elevated barrier uptake at baseline greater than 2 standard deviations of a healthy reference cohort | Up to 12 months
  Time to acute exacerbation or respiratory hospitalization will be an aggregate value and will be recorded in months
Time to acute exacerbation or respiratory hospitalization in individuals with decreased RBC transfer at baseline, lower than 2 standard deviations of a healthy reference cohort | Up to 12 months
  Time to acute exacerbation or respiratory hospitalization will be an aggregate value and will be recorded in months

CONTACTS AND LOCATIONS:
Overall Officials: Robert M Tighe, MD, Principal Investigator — Duke University Health Systems
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No